CLINICAL TRIAL: NCT05085093
Title: Protective Efficacy of HPV Vaccination After Treatment of HPV Related Diseases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20212121
Record Dates: First submitted 2021-10-17; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: HPV Vaccination、HPV Related Diseases、Protective Efficacy
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: HPV vaccine group
  Interventions: Biological: HPV vaccine
- Control group: non HPV vaccine group

INTERVENTIONS:
Biological: HPV vaccine — Patients choose to be vaccinated or not to be vaccinated with HPV vaccine according to their own wishes
  Groups: Study Group

SUMMARY:
To understand the HPV infection status and subtype distribution of patients, and to study the protective effect of prophylactic HPV vaccination on the recurrence of HPV related diseases after treatment through a prospective cohort study. To provide data support for the primary prevention of HPV related diseases in Chinese women after treatment, and to analyze the related factors of HPV related disease recurrence and HPV continuous positive.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women aged 18-45, of childbearing age or before perimenopause (patients without pregnancy plan within two years); 2. Patients diagnosed as condyloma acuminatum, vaginal intraepithelial lesions (high-grade and low-grade lesions), cervical intraepithelial lesions (high-grade and low-grade lesions), vulvar intraepithelial lesions (high-grade and low-grade lesions), cervical cancer (IA1-IIA2 stage) and treated within 3 months; 3. No surgical contraindications such as severe center of heart, lung and other organ dysfunction and abnormal hemagglutination; 4. Fully know the treatment method, sign informed consent, and actively cooperate with follow-up.

Exclusion Criteria:

* 1. Participating in other clinical trials; 2. Use immunoglobulin or blood products within 3 months before vaccination; 3. Hypersensitivity to vaccine active ingredients or any dressing ingredients; 4. Acute stage of moderate and severe diseases; 5. Acute stage of severe immune deficiency diseases and autoimmune diseases; 6. Pregnant women and lactating patients; 7. Patients with planned pregnancy within 2 years; 8. Less than 18 years old and more than 45 years old.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — The diseases in this study mainly occurred in female groups
Study Population: All patients with HPV related diseases
Sampling Method: Probability Sample
Enrollment: 414 (Estimated)
Dates: Start 2021-09-18 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
recurrence | 6 months after operation
  If The lesions were found again more than 6 months after operation (pathological diagnosis)
Persistent HPV infection | At least 12 months
  At least 12 months apart, cervical vaginal / external genital swabs or tissue biopsies were taken for 2 or more consecutive times, and HPV detection and analysis showed that the same HPV type was positive

CONTACTS AND LOCATIONS:
Overall Officials: hong Yang, professional, Study Chair — The First Affiliated Hospital，Air Force Medical University,Xi'an, Shaanxi, China
Locations (1):
- The First Affiliated Hospital, Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
We haven't decided whether to share the data yet